CLINICAL TRIAL: NCT00322842
Title: Treatment With AMD3100 in Non-Hodgkin's Lymphoma and Multiple Myeloma Patients to Increase the Number of Peripheral Blood Stem Cells When Given a Mobilizing Regimen of G-CSF
Brief Title: Treatment With AMD3100 (Plerixafor) in Non-Hodgkin's Lymphoma and Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: AnorMED (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMD3100-EU21
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Results first posted 2010-11-25 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-02

CONDITIONS: Lymphoma, Non-Hodgkin; Multiple Myeloma
Keywords: Non-Hodgkin's lymphoma; Multiple Myeloma; Stem cell mobilization
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — Granulocyte Colony-Stimulating Factor; plerixafor

ARMS (2):
- Non-Hodgkin's Lymphoma (NHL) (Experimental): Participants with NHL were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor
- Multiple Myeloma (MM) (Experimental): Participants with MM were mobilized with granulocyte colony-stimulating factor (G-CSF) 10 µg/kg/day for 4 days. Plerixafor 240 µg/kg was given the evening of day 4 and G-CSF given the next morning followed by apheresis. Evening doses of plerixafor and morning doses of G-CSF followed by apheresis continued for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Interventions: Drug: G-CSF Plus Plerixafor

INTERVENTIONS:
Drug: G-CSF Plus Plerixafor — Participants underwent mobilization with G-CSF 10 µg/kg/day for 4 days, administered by subcutaneous injection (SC) injection each morning. On the evening of Day 4, participants received a dose of plerixafor 240 µg/kg, administered by SC injection. On Day 5, participants returned to the clinic and received a morning dose of G-CSF 10 µg/kg and underwent apheresis approximately 10 to 11 hours after the dose of plerixafor (within 60 minutes after administration of G-CSF). Participants continued to receive an evening dose of plerixafor followed the next day by a morning dose of G-CSF and apheresis for up to a maximum of 5 aphereses or until ≥ 5*10^6 CD34+ cells/kg were collected.
  Other Names: Mozobil; AMD3100

SUMMARY:
This study evaluates the safety of plerixafor and other outcomes that are purely exploratory in nature. One other pre-specified outcome is to evaluate an interval of 10-11 hours between dosing with plerixafor and the beginning of apheresis to determine if there will be at least a 2-fold increase in circulating CD34+ cells. Data from this protocol will assist in the determination of the dosing schedule for future studies.

DETAILED DESCRIPTION:
Participants with non-Hodgkin's lymphoma and multiple myeloma who have undergone prior cyto-reductive chemotherapy and are to be autologously transplanted will be treated with a combination of plerixafor and granulocyte colony-stimulating factor (G-CSF) mobilization regimen on the day prior to apheresis. The only change to standard of European care is the addition of plerixafor to a G-CSF mobilizing regimen. Participants will undergo mobilization with G-CSF (10 µg/kg each day) and on each day prior to apheresis will receive plerixafor (240 µg/kg). Participants will undergo apheresis for up to 5 consecutive days in order to collect the target number of (≥ 5*10^6) CD34+ stem cells/kg. Participants will be transplanted with cells obtained from the G-CSF and plerixafor mobilization regimen. The number of CD34+ cells mobilized in the peripheral blood from the time of the plerixafor dose to just prior to apheresis and those harvested in the apheresis product will be measured. The number of apheresis sessions required to obtain ≥ 5*10^6 CD34+ cells/kg will also be measured. Success of the transplantation(s) will be evaluated by the time to engraftment of poly-morphonuclear leukocytes (PMN) and platelets (PLT). Participants will be followed for durability of their transplant for 12 months following transplantation.

This study was previously posted by AnorMED, Inc. In November 2006, AnorMED, Inc. was acquired by Genzyme Corporation. Genzyme Corporation is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-Hodgkin's lymphoma (NHL) or multiple myoloma (MM) eligible for autologous transplantation
* No more than 3 prior regimens of chemotherapy
* More than 4 weeks since last cycle of chemotherapy. Patient recovered from all acute toxic effects of prior chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* White blood cell (WBC) count >3.0*10^9/L
* Absolute polymorphonuclear cells (PMN) count >1.5*10^9/L
* Platelet (PLT) count >100*10^9/L
* Serum creatinine <=2.2 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT) and total bilirubin <2 x upper limit of normal (ULN)
* Left ventricle ejection fraction >45% by normal echocardiogram or multiple-gated acquisition (MUGA) scan
* Negative for human immunodeficiency virus (HIV)
* Women of child bearing potential who agreed to use an approved form of contraception.

Exclusion Criteria:

* Patients who have failed previous collections
* Brain metastases or carcinomatous meningitis
* History of ventricular arrhythmias
* History of paresthesias
* A co-morbid condition which, in the view of the investigator, renders the patient at high risk for treatment complications
* A residual acute medical condition resulting from prior chemotherapy
* Acute infection
* Fever (temp >38°C/100.4°F)
* Patients whose actual body weight exceeds 150% of their ideal body weight
* Patients who previously received experimental therapy within 4 weeks of enrolling in this study or who are currently enrolled in another experimental study during the mobilization period
* Positive pregnancy test in female patients
* Lactating females
* Patients of child-bearing potential unwilling to implement adequate birth control.
* Patients who have deterioration of their clinical status or laboratory parameters between the time of enrolment and transplant (such that they no longer meet entry criteria) may be removed from study at the discretion of the treating physician, principal investigator, or sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (3):
- Germany (3):
  - University of Cologne, Cologne
  - Carl Gustav Carus University Hospital, Dresden
  - University of Heidelberg, Heidelberg

REFERENCES:
- [Background] Fruehauf S, Seeger T, Maier P, Li L, Weinhardt S, Laufs S, Wagner W, Eckstein V, Bridger G, Calandra G, Wenz F, Zeller WJ, Goldschmidt H, Ho AD. The CXCR4 antagonist AMD3100 releases a subset of G-CSF-primed peripheral blood progenitor cells with specific gene expression characteristics. Exp Hematol. 2006 Aug;34(8):1052-9. doi: 10.1016/j.exphem.2006.06.003. PMID 16863911
- [Result] Fruehauf S, Ehninger G, Hubel K, Topaly J, Goldschmidt H, Ho AD, Muller S, Moos M, Badel K, Calandra G. Mobilization of peripheral blood stem cells for autologous transplant in non-Hodgkin's lymphoma and multiple myeloma patients by plerixafor and G-CSF and detection of tumor cell mobilization by PCR in multiple myeloma patients. Bone Marrow Transplant. 2010 Feb;45(2):269-75. doi: 10.1038/bmt.2009.142. Epub 2009 Jul 13. PMID 19597422
- [Result] Fruehauf S, Veldwijk MR, Seeger T, Schubert M, Laufs S, Topaly J, Wuchter P, Dillmann F, Eckstein V, Wenz F, Goldschmidt H, Ho AD, Calandra G. A combination of granulocyte-colony-stimulating factor (G-CSF) and plerixafor mobilizes more primitive peripheral blood progenitor cells than G-CSF alone: results of a European phase II study. Cytotherapy. 2009;11(8):992-1001. doi: 10.3109/14653240903121245. PMID 19929463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Started | 4 | 31
Completed | 2 (One participant discontinued (d/c) treatment early, received a transplant, and completed the study.) | 29 (One participant d/c treatment early, received a transplant, and was lost to follow-up after 6 months)
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Refused transplant | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | Total
Number analyzed (Participants) | 4 | 31 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.1) | 58.8 (7.3) | 58.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 1 | 19 | 20
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4 | 30 | 34
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Overall Safety Summary of Treatment Emergent Adverse Events (TEAE)
Description: Number of participants with treatment emergent adverse events (TEAEs) collected from Day 1 (start of G-CSF mobilization) to the day before starting chemotherapy (approximately day 38). AEs were graded by the investigator using the World Health Organization (WHO) Adverse Event Grading Scale and were assessed for severity (mild, moderate, severe) and relatedness to study treatment (5 step scale from 'not related' to 'definitely related').
Time Frame: Day 1 to approximately Day 38 (before start of chemotherapy)
Population: Safety population - all participants who received at least 1 dose of plerixafor.
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 4 | 31 | 35
participants
  Participants reporting ≥ 1 AE | 4 | 20 | 24
  AE Severity (Mild) | 2 | 16 | 18
  AE Severity (Moderate) | 2 | 4 | 6
  AE Severity (Severe) | 0 | 0 | 0
  AE Relationship to Drug (Not Related) | 4 | 18 | 22
  AE Relationship to Drug (Probably Not Related) | 0 | 0 | 0
  AE Relationship to Drug (Possibly Related) | 0 | 2 | 2
  AE Relationship to Drug (Probably Related) | 0 | 0 | 0
  AE Relationship to Drug (Definitely Related) | 0 | 0 | 0

2. Secondary Outcome: Fold (i.e., Relative) Increase in Peripheral Blood (PB) CD34+ Cells/µL After First Dose of Plerixafor
Description: The fold increase was measured using local lab values and is the ratio of post first dose (pre-apheresis) PB CD34+ cells/µL)/pre-plerixafor dosing PB CD34+ cells/µL)
Time Frame: Days 4-5 (first dose of plerixafor to apheresis)
Population: Intent to treat population
Measure: Median (Full Range); unit: ratio
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 4 | 31 | 35
ratio | 2.6 (1.2) [2.0 to 4.7] | 2.6 (1.4) [1.1 to 6.9] | 2.6 (1.3) [1.1 to 6.9]

3. Other Pre Specified Outcome: Median Cumulative Number of CD34+ Cells Collected During Apheresis
Description: Median total number of CD34+ cells collected during apheresis as measured by a central lab.
Time Frame: Days 5-8
Population: Intent to treat population. Samples from two participants were not analyzed by the central lab.
Measure: Median (Full Range); unit: CD34+ cells (*10^6 / kg)
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 4 | 29 | 35
CD34+ cells (*10^6 / kg) | 8.3 [4.9 to 17.6] | 7.1 [0.1 to 35.7] | 7.4 [0.1 to 35.7]

4. Secondary Outcome: Number of Transplants in Which Participants Achieved Polymorphonuclear Leukocyte (PMN) Engraftment by Day 12 But No Later Than Day 21 Post Peripheral Blood Stem Cell (PBSC) Transplant
Description: Participants were monitored for polymorphonuclear leukocyte (PMN) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: Participants who had transplants. Fifteen participants had tandem transplants. The date of initial PMN engraftment was missing for 11 transplants, which were later shown to have durable grafts.
Measure: Number; unit: number of transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 3 | 30 | 33
Number analyzed (transplants) | 3 | 45 | 48
number of transplants
  ≤ Day 12 | 0 | 8 | 8
  Day 13 to Day 21 | 2 | 25 | 27
  ≥ Day 22 | 1 | 1 | 2
  Unknown | 0 | 11 | 11

5. Other Pre Specified Outcome: Number of Transplants in Which Participants Achieved Platelet (PLT) Engraftment by Day 12 But No Later Than Day 21 Post Peripheral Blood Stem Cell (PBSC) Transplant
Description: Participants were monitored for platelet (PLT) engraftment as per the local standard of care. The target for engraftment was 12 days after PBSC transplant and no transplant taking longer than 21 days for engraftment.
Time Frame: 2 months
Population: Participants who had transplants. Fifteen participants had tandem transplants.
Measure: Number; unit: number of transplants
Units Other Than Participants: transplants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 3 | 30 | 33
Number analyzed (transplants) | 3 | 45 | 48
number of transplants
  ≤ Day 12 | 0 | 32 | 32
  Day 13 to Day 21 | 2 | 13 | 15
  ≥ Day 22 | 1 | 0 | 1

6. Other Pre Specified Outcome: Number of Participants With Durable Engraftment 12 Months After Transplantation
Description: The number of participants maintaining a durable graft 12 months after autologous transplantation. A durable graft is defined as the maintenance of normal blood counts.
Time Frame: Approximately 13 months (12 months post-transplant )
Population: Participants who had transplants and engraftment data 12 months after transplantation
Measure: Number; unit: participants
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 2 | 29 | 31
participants | 2 | 29 | 31

7. Secondary Outcome: Increase in Peripheral Blood (PB) CD34+ Cells From Steady-state Hematopoiesis to Pre-leukapheresis in G-CSF+Plerixafor Treated Participants Compared to Historical Controls Treated With G-CSF Alone or Chemotherapy and G-CSF
Description: A comparison of the effectiveness in mobilizing peripheral blood CD34+ cells between this study's treatment regimen (G-CSF plus plerixafor) to other treatment options: G-CSF alone, and chemotherapy with G-CSF.
Time Frame: up to day 8
Population: Analysis was not performed. Historical data was not available.
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM) | All Participants
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First day of G-CSF administration to the day prior to chemotherapy/ablative treatment in preparation of first transplant. This period includes the G-CSF, plerixafor treatment and rest period.
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. Each AE table includes events, regardless of reported relationship to study treatment or grade.
Arm/Group | Non-Hodgkin's Lymphoma (NHL) | Multiple Myeloma (MM)
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/31
Other Adverse Events (participants affected / at risk) | 4/4 | 20/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=4) | Multiple Myeloma (MM) (N=31)
Pyrexia (General disorders) | 1 | 0
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Hodgkin's Lymphoma (NHL) (N=4) | Multiple Myeloma (MM) (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Asthenia (General disorders) | 1 | 0
Catheter site pain (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Bacterial infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Hypertonia (Nervous system disorders) | 0 | 1 — Medical review concluded that this event, which was not related to study drug, would have been more appropriately coded to hypertension.
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1 — Medical review concluded that this event, which was not related to study drug, would have been more appropriately coded to hypotension.
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 2
Renal pain (Renal and urinary disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiovascular insufficiency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.